CLINICAL TRIAL: NCT06467500
Title: A Prospective, Open-label, Single-center, Single-arm Phase II Clinical Study of Cadonilimab (AK104) Combined With Monotherapy Chemotherapy in Patients With Advanced Non-small Cell Lung Cancer (NSCLC) With Negative Driver Genes and Failed Immunotherapy
Brief Title: A Prospective, Open-label, Single-center, Single-arm Phase II Clinical Study of Cadonilimab (AK104) Combined With Monotherapy Chemotherapy in Patients With Advanced Non-small Cell Lung Cancer With Negative Driver Genes and Failed Immunotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xin-Hua Xu (Other)
Responsible Party: Sponsor-Investigator, Xin-Hua Xu, professor, China Three Gorges University, Yichang, China
Organization: China Three Gorges University, Yichang, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTGU010
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bispecific antibody plus Chemotherapy (Experimental)
  Interventions: Drug: Cadonilimab (AK104)

INTERVENTIONS:
Drug: Cadonilimab (AK104) — Subjects participated in a study where they received cadonilimab intravenously at 6mg/kg every two weeks, prepared in 100mL of normal saline (0.9% NaCl), with a final concentration range of 0.2-5.0mg/mL. The infusion solution must be used within 4 hours of preparation. Treatment continued until disease progression (PD), unacceptable toxicity, or 24 months, whichever came first. Patients who investigators deemed could still benefit from cadonilimab post-PD were allowed continued treatment. Chemotherapy regimens were selected by investigators based on prior medication use, including gemcitabine, pemetrexed, docetaxel, albumin-bound paclitaxel, or vinorelbine as second- or third-line therapy

SUMMARY:
The aim of evaluating the efficacy and safety of cadonilimab combined with monotherapy chemotherapy in patients with advanced non-small cell lung cancer (NSCLC) with negative driver genes who have failed previous immunotherapy is to provide a more effective and safe treatment option for these patients.

DETAILED DESCRIPTION:
Cadonilimab (AK104), China's first globally developed bispecific antibody targeting both PD-1 and CTLA-4, has demonstrated manageable safety and promising anti-tumor activity in female cervical cancer, esophageal squamous cell carcinoma, and hepatocellular carcinoma. However, there is currently no available data on the efficacy and safety of cadonilimab combined with monotherapy chemotherapy for treating advanced non-small cell lung cancer (NSCLC) with negative driver genes and previous immunotherapy failure. Therefore, this study aims to prospectively and openly evaluate the efficacy and safety of cadonilimab combined with monotherapy chemotherapy in treating patients with advanced NSCLC with negative driver genes and previous immunotherapy failure using a single-arm trial design. The goal is to provide a more effective and safe treatment option for these patients.

ELIGIBILITY:
Inclusion Criteria:

Voluntarily participate in clinical research; Fully understand and be informed of this study and sign the informed consent form;

1. Age ≥ 18 and ≤ 75, male or female;
2. ECOG physical performance score of 0-2;
3. Patients with histologically confirmed squamous or non-squamous advanced non- small cell lung cancer (according to AJCC, 8th edition);
4. Patients who tested negative for driver genes after genetic testing;
5. Patients who have undergone previous systemic therapy and failed anti-PD-1/PD- L1 immunotherapy;
6. Presence of at least one measurable lesion as defined by Recist criteria 1.1;
7. Liver function: Total serum bilirubin ≤ 1.5 × ULN; For subjects without liver metastasis, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN, and for those with liver metastasis, ALT and AST ≤ 5 × ULN;
8. Renal function: Serum creatinine ≤ 1.5 × ULN or creatinine clearance rate ≥ 45 mL/min (using the Cockcroft/Gault formula); Blood routine: Absolute neutrophil count ≥ 1.5 × 109/L, platelet count ≥ 70 × 109/L; Hemoglobin ≥ 80g/L (no blood transfusion or use of hematopoietic stimulating drugs for correction within 7 days before screening) with an expected lifespan of more than 3 months.

Exclusion Criteria:

1. ECOG physical performance score > 2;
2. Previous treatment with bispecific antibodies;
3. Participation in other clinical trials within 30 days prior to screening;
4. Tumor metastasis to the brain and/or leptomeninges;
5. History of other malignancies (excluding cervical carcinoma in situ or skin basal cell carcinoma that has been cured, and other malignancies that have been cured for more than 5 years);
6. Accompanied by other serious diseases, including but not limited to:

   1. Difficult-to-control congestive heart failure (NYHA class III or IV), unstable angina, poorly controlled arrhythmia, uncontrolled moderate to severe hypertension (SBP > 160mmHg or DBP > 100mmHg);
   2. Severe active infection;
   3. Difficult-to-control diabetes (referring to large fluctuations in blood sugar despite standard insulin therapy and frequent blood glucose monitoring, affecting the patient's life and frequently causing hypotension);
   4. Mental illness affecting informed consent and/or protocol compliance.
7. Allergy to the drugs used in this protocol or their ingredients;
8. Pregnant (confirmed by blood or urine HCG testing) or breastfeeding women, or subjects of reproductive age who are unwilling or unable to take effective contraceptive measures (applicable to both male and female subjects) until at least 6 months after the last experimental treatment;
9. Investigators consider it inappropriate to participate in this study;
10. Unwilling to participate in this study or unable to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | approximately 24 months
  The objective response rate (ORR) refers to the proportion of patients whose tumor shrinks by a certain percentage (generally 30%) and maintains this reduction for a certain period of time (generally 4 weeks).

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | approximately 24 months
  Disease Control Rate (DCR) is defined as the proportion of patients with a cancer or tumor who experience a reduction in the size of the disease, no progression of the disease, or stable disease conditions for a specified period of time after receiving a particular treatment. This typically includes patients who achieve complete response (CR), partial response (PR), or stable disease (SD).
Duration of Response (DoR) | approximately 24 months
  Duration of Response (DoR), which stands for Duration of Response, refers to the length of time from the point when a subject achieves a confirmed complete response (CR) or partial response (PR) to the time when the first sign of disease progression or death due to any cause occurs.
Progression-free survival (PFS) | approximately 24 months
  PFS was defined as the time between the date of randomization and the date of first documented disease progression or death, whichever occurs first. Disease progression was determined based on investigator assessment using response evaluation criteria In solid tumors (RECIST) v1.1.
Overall Survival (OS) | approximately 24 months
  Overall Survival (OS) was defined as the time from the date of randomization to the date of death due to any cause.Data for participants who were not reported as dead at the time of analysis was censored at the date when they were last known to be alive.
Adverse event (AE) | approximately 24 months
  Adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Central Hospital of Yichang City, the First Clinical Medical College of Three Gorges University, Yichang, China